CLINICAL TRIAL: NCT05902052
Title: Master of Science, Registery Nurse
Brief Title: Development of Open Heart Surgery Patient Care Protocol and Its Effect on Post-sternotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Lecturer, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0001
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result; Pain, Postoperative; Nursing Caries
Keywords: Heart Surgery; pain; sternotomy; protocol; nursing
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — CARE protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Heart Surgery Patient Care Protocol (Experimental): Specific Practices for Pain in the Protocol
  * Evaluation of patients' pain in the extubated period with the Visual Anolog Scale
  * Active participation of the patient in pain reporting
  * Regular questioning of the patient's pain
  * Questioning pain at rest and movement
  * Implementing nursing interventions in painful condition (VAS≤ 4)
  Interventions: Other: Care Protocol
- Standart Care Protocol (No Intervention): Standard care of intensive care will be given.

INTERVENTIONS:
Other: Care Protocol — Evaluation of patients' pain in the extubated period with the Visual Anolog Scale Active participation of the patient in pain reporting Regular questioning of the patient's pain Questioning pain at rest and movement Implementing nursing interventions in painful condition (VAS≤ 4)
  Arms: Open Heart Surgery Patient Care Protocol

SUMMARY:
Open heart surgery method is generally used in the treatment of cardiovascular diseases. Sternotomy is the process of opening the sternum. After sternotomy, individuals experience ongoing pain in the anterior thorax. Despite developing pain methods and treatments, individuals undergoing cardiovascular surgery suffer from pain that cannot be managed well. Patients undergoing cardiac surgery experience severe pain for the first 48 hours and are in intensive care during this period. Pain is the most important stress factor for intensive care patients. The nurse and health care team should play a key role and take an active role in the management and evaluation of pain. However, there are not enough studies trying to define the role of the nurse in the management of postoperative pain. Protocols are used to provide pain management and routine pain assessment in intensive care units. The use of protocols provides maximum care to the patient, while reducing the cost. It also ensures the patient's participation in the treatment. While protocols ensure that practices are converted into evidence-based ones, they also prevent disruptions in treatment. As a result, management of the pain experiences of patients with sternotomy who underwent open heart surgery in the intensive care unit with the developed protocol; It will guide the improvement and development of pain management. It is thought that the protocol will address the pain of individuals undergoing open heart surgery in a holistic way. In addition, no study has been found in the literature that includes the development of a protocol for the pain of intensive care patients undergoing open heart surgery. For this reason, it is thought that the study will shed light on the literature by being a resource in the management and improvement of pain.

DETAILED DESCRIPTION:
In this study, it is aimed to develop the open heart surgery patient care protocol and to examine its effect on the pain that develops after sternotomy. The research is planned to be carried out on the patients in the Cardiovascular Surgery Intensive Care Unit of Research Hospital. The sample size of this study was decided by power analysis. The G-Power statistics program is based on Type 1 error 0.05 and 80% power. In the power analysis of Akbayrak and Tosun's (2002) thesis study, using the results showing the average score of the satisfaction level of the patients with and without the care protocol, the sample size was determined as 17 patients for each group and 34 patients in total. However, in order to meet the parametric test assumptions, it was decided to include at least 30 people in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sternotomy who underwent Coronary Artery Bypass Graft surgery,
* Patient with sternotomy who underwent valve surgery,
* Being 18 years or older,
* Volunteering to participate in the research,
* Being at a level to adequately answer the questions asked cognitively,
* Experiencing pain at least once after the surgery,
* No complications (unable to wean from mechanical ventilator support, inability to discontinue inotropic support) until the period of transfer to the postoperative service.

Exclusion Criteria:

* Desiring to leave the study group during the conduct of the research,
* Delirium development in the patient during the conduct of the study,
* The patient for whom emergency surgery has been decided.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 days
  Visual Analog Scale
Scale for Evaluation of the Quality of Care Given to the Patient in Relief of Postoperative Pain | Just before being transferred to intensive care
  The scale consists of 14 items and has 3 sub-dimensions related to nursing interventions, pain management and environment. Likert type scale was used in the evaluation. 1 means "strongly disagree" and 5 means "strongly agree". The scale Cronbach's coefficient was 0.81 and the main score obtained from the scale was 45.8 ± 10.8. The scale is a reliable and valid instrument in Turkish language.
Analgesic use | 3 days
  Number of analgesic use
Type of analgesic | 3 days
  Type of analgesic

SECONDARY OUTCOMES:
Anxiety | Before going into surgery, Just before being transferred to intensive care
  State Anxiety Scale The scale consists of a total of 20 items and each item is evaluated as (1) none, (2) a little, (3) a lot, (4) completely. There are direct and reversed statements in the scale. Positive emotions are defined by inverted statements, and those with a weight of 1 turn into a 4 in a rating, and a weight of 4 turns into a 1. In reversed statements, answers with a value of 1 indicate high anxiety, and those with a value of 4 indicate low anxiety. The total score of the reversed statements is subtracted from the calculated direct statement score, and the unchanged value 50 is added to the resulting number. The total score is between 20-80. According to the score calculated on the scale, 0-19 means no anxiety, 20-39 means mild, 40-59 moderate, 60-79 high anxiety.
Blood pressure | 3 days
  Measuring arterial blood pressure Systolic blood pressure (the first and higher number) measures pressure inside your arteries when the heart beats.
  Diastolic blood pressure (the second and lower number) measures the pressure inside the artery when the heart rests between beats.
respiratory | 3 days
  respiratory rate
Fever | 3 days
  Temperature measurement. A fever is a body temperature that is higher than normal. A normal temperature can vary from person to person, but it is usually around 98.6 °F (37 °C).
Heart rate | 3 days
  Heart rate measurement. A normal resting heart rate for adults ranges from 60 to 100 beats per minute.
Oxygen Saturation | 3 days
  Oxygen saturation can be measured using a pulse oximetry device, which is a non-invasive method to measure arterial oxygen saturation level. A pulse oximeter can measure oxygen saturation. It is a noninvasive device placed over a person's finger. It measures light wavelengths to determine the ratio of the current levels of oxygenated hemoglobin to deoxygenated hemoglobin. The use of pulse oximetry has become a standard of care in medicine.
Partial pressure of carbon dioxide | 3 days
  Blood gases are a measurement of how much oxygen and carbon dioxide are in your blood. They also determine the acidity (pH) of your blood. The partial pressure of carbon dioxide (PCO2) is the measure of carbon dioxide within arterial or venous blood. It often serves as a marker of sufficient alveolar ventilation within the lungs. Generally, under normal physiologic conditions, the value of PCO2 ranges between 35 to 45 mmHg, or 4.7 to 6.0 kPa.
Partial pressure of oxygen | 3 days
  Blood gases are a measurement of how much oxygen and carbon dioxide are in your blood. They also determine the acidity (pH) of your blood.Partial pressure of oxygen (PaO2): 75 to 100 millimeters of mercury (mm Hg), or 10.5 to 13.5 kilopascal (kPa)

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Atatürk Training and research hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No